CLINICAL TRIAL: NCT00864773
Title: Intraocular Concentrations of Growth Factors and Cytokines in Chronic Central Serous Chorioretinopathy And the Effect of Therapy With Bevacizumab
Brief Title: The Effect of Therapy With Bevacizumab in Chronic Central Serous Chorioretinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Hallym University Medical Center, Hallym University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009-3-16
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2009-03-19 (Estimated); Status verified 2009-03

CONDITIONS: Central Serous Chorioretinopathy
MeSH Terms: conditions — Central Serous Chorioretinopathy | interventions — Intravitreal Injections; Bevacizumab

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: intravitreal injection with anterior paracentesis — 0.1cc Aqueous humor samples were taken each time an intravitreal injection of bevacizumab (2.5 mg in 0.1 ml)
  Other Names: Bevacizumab (Avastin, Genetech); an antibody to vascular endothelial growth factor (VEGF)

SUMMARY:
The pathophysiology of central serous chorioretinopathy remains controversial. traditional treatment is laser photocoagulation or photodynamic therapy.Recently Bevacizumab (Avastin, Genetech),an antibody to vascular endothelial growth factor (VEGF),has known antipermeability properties and therefore may theoretically reverse the changes seen in central serous chorioretinopathy. The aim of this study is To investigate concentrations of growth factors and inflammatory cytokines and to report the effect of therapy with bevacizumab in eyes with central serous chorioretinopathy

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of central serous chorioretinopathy
* Idiopathic neurosensory retinal elevation demonstrated by optical coherent tomography
* Presence of focal leaks at the level of the RPE on fluorescein angiography

Exclusion Criteria:

* Known side effects of systemic bevacizumab administration
* Have a significant cardiovascular or thromboembolic history or were pregnant

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Concentrations of growth factors and inflammatory cytokines in Aqueous humor | at baseline

SECONDARY OUTCOMES:
Central macular thickness at optical coherence tomography | baseline, 1 month, 3 months, 6 months